CLINICAL TRIAL: NCT00208611
Title: Assessment of Cobalamin Status and Responses to Supplementation in Patients With Parkinson's Disease : a Pilot Study
Brief Title: Vitamin B12 Status and Response to Vitamin B12 Supplementation in Patients With Parkinson's Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding ended and enrollment not completed within a certain time period
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Marian L. Evatt, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple
Other Study IDs: IRB00045854
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label Treatment (Experimental): Levodopa-treated Parkinson's Disease subjects with vitamin B12 < 200 pg/ml given oral vitamin B12 supplement
  Interventions: Dietary Supplement: Vitamin B12 Supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin B12 Supplementation — 1000 micrograms daily
  Other Names: vitamin B12

SUMMARY:
Based on Parkinson's disease (PD)/vitamin B12 deficiency symptom overlap and PD patients' propensity to avoid protein (the dietary source of vitamin B12), this study proposes to prospectively investigate the vitamin B12 status of PD patients over time. In addition, this study will provide critical pilot data evaluating the efficacy of treating those patients considered to have below-normal vitamin B12 levels in serum. Further, it will also explore the concept that supplementing PD patients having "low-normal" vitamin B12 levels with vitamin B12 improves either the non-motor PD symptoms or homocysteine levels in PD patients receiving levodopa.

Study Hypotheses:

1. Serum cobalamin (B12) concentrations in patients with Parkinson's disease (PD) are significantly lower than B12 concentrations in a) cohabiting spousal caregiver controls; and b) population-based, age-matched controls.
2. Supplementation with B12 in levodopa-treated PD patients with low (<200 pg/ml) or low-normal (200-300 pg/ml) serum B12 levels is associated with significant improvement in their non-motor symptoms and reduces total plasma homocysteine concentration [Hcy], a known biomarker for risk of dementia and cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in Emory Healthcare System at least once between 1/1/2002 and 05/31/2006 with idiopathic Parkinson's disease (defined as):
* >2 of cardinal signs/symptoms of Parkinson's disease (bradykinesia, tremor, rigidity)
* >50% improvement of symptoms when dopaminergic therapy started
* Cohabiting spousal caregivers (without Parkinson's disease) of patients enrolled in study are also eligible (but not required) to participate

  * Coexisting depression, if present, is stable
  * Normal thyroid screen (done at Screening Visit or at Emory Healthcare System within 3 months of Screening Visit)
  * Males must have normal fasting testosterone levels (done at Screening visit or within 6 months of Screening Visit)

Exclusion Criteria:

* Unstable medical conditions (terminal cancer, angina, etc) which could interfere with study assessments or put patient at risk for not completing the assessments.
* Dopaminergic-unresponsive parkinsonism (i.e., patient has suspected multiple systems atrophy (MSA), vascular or another form of parkinsonism)
* Prior history of vitamin B12 deficiency or taking vitamin B12 supplements or injections (single multivitamin supplements are not an exclusion criteria)
* Untreated testosterone or thyroid abnormality

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Vitamin B12 concentration | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marian L Evatt, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States